CLINICAL TRIAL: NCT04809311
Title: Fully Decentralised Clinical Study Exploring Remote Collection of Glycaemic and Behaviometric Data Among Participants With Type 2 Diabetes Mellitus on Different Treatment Regimens
Brief Title: Remote Study Collecting Blood Glucose Values and Activity Data in Patients With Type 2 Diabetes on Different Treatments
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1535-7774; U1111-1254-5030 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Other oral antidiabetic drugs (OADs) ± metformin: Patients will continue their antidiabetic treatment as per usual clinical practice at the discretion of their own treating physician
  Interventions: Drug: Oral antidiabetetic drugs
- Basal insulin ± OADs: Patients will continue their antidiabetic treatment as per usual clinical practice at the discretion of their own treating physician
  Interventions: Drug: Basal insulin
- Glucagon-like peptide-1 (GLP-1) ± Basal insulin (loose and fixed combination) ± OADs: Patients will continue their antidiabetic treatment as per usual clinical practice at the discretion of their own treating physician
  Interventions: Drug: Basal insulin; Drug: Glucagon-like peptide-1 (GLP-1)

INTERVENTIONS:
Drug: Oral antidiabetetic drugs — During the study, no medical drugs will be supplied to the patients. Patients will continue their antidiabetic treatment independently of this study and at the treating physician's discretion as part of usual clinical practice.
  Approximately 12-week study duration
  Groups: Other oral antidiabetic drugs (OADs) ± metformin
Drug: Basal insulin — During the study, no medical drugs will be supplied to the patients. Patients will continue their antidiabetic treatment independently of this study and at the treating physician's discretion as part of usual clinical practice.
  Approximately 12-week study duration
  Groups: Basal insulin ± OADs; Glucagon-like peptide-1 (GLP-1) ± Basal insulin (loose and fixed combination) ± OADs
Drug: Glucagon-like peptide-1 (GLP-1) — During the study, no medical drugs will be supplied to the patients. Patients will continue their antidiabetic treatment independently of this study and at the treating physician's discretion as part of usual clinical practice.
  Approximately 12-week study duration
  Groups: Glucagon-like peptide-1 (GLP-1) ± Basal insulin (loose and fixed combination) ± OADs

SUMMARY:
Earlier protocol ID was NN1250-4630, protocol ID is changed to NN1535-7774. The purpose of this study is to collect blood glucose values and activity data in patients with type 2 diabetes for approximately 12 weeks using electronic devices in a full virtual clinical setting. Virtual clinical setting means that all data are collected by use of participants' personal smartphone and study-related apps. In other words, everything will be handled without any visits to a hospital or doctor.

For collection of participants' blood glucose values participants will receive two different blood glucose monitors. One where participants cannot see the blood glucose values and one where participants can see the blood glucose values. Participants must wear them consecutively for 2 and 10 weeks, respectively. Further, participants will be asked to self-apply the monitors on their upper arm.

For collection of participants' activity data participants will receive an activity tracker, which participants will wear on the wrist throughout the study.

The study does not include any study medication and participants will continue the current antidiabetic treatment as prescribed to participants by their own physician. If any questions about the treatment and/or health condition while participating in the trial, participants should consult your own physician If participants are in doubt about what the blood glucose values mean or whether participants should react to the blood glucose values, participants need to contact the research staff or their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to consent via the e-consent process before any study-related activities takes place (study-related activities are any procedure related to recording of data according to the protocol)
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Diagnosed T2DM for more than 3 months prior to signing the informed consent
* On one of the following treatments for T2DM:

  1. Metformin ± other OADs
  2. Basal insulin ± OADs
  3. GLP-1 ± Basal insulin (loose and fixed combination) ± OADs
* Willingness to, and capable of applying and using the study devices
* Willingness to follow study procedures
* Fluent in Danish both oral, reading and in writing
* In possession of a compatible smartphone throughout the study, meaning that the smartphone fulfils the criteria to the operating system for using the devices needed for the study

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Participation in any other study investigating diabetes.
* Patients who do not have a blood glucose meter at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus on different treatment regimens.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Participant invited to consent and consented via e-signature (Yes/No) | During Screening (Week -2 to week 0 )
  Measured as count of participants.
Participant with at least 70% unblinded CGM (continuous glucose monitoring) data (Yes/No) | From time of first unblinded CGM measurement until 10 weeks after the time of first unblinded CGM measurement
  Measured as Count of participants.
Participant completion of questionnaires and per protocol planned remote visits (RVs) | From week 0 until end of study (week 12)
  % of questionnaires and RVs completed.

SECONDARY OUTCOMES:
Time in range (TIR) (3.9-10 mmol/L) | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
  % of time.
Time above range (TAR) (above 10 mmol/L) | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
  % of time.
Time below range (TBR) L1 (3.0-3.9 mmol/L) | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
  % of time.
Time below range (TBR) L2 (below 3.0 mmol/L) | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
  % of time.
Mean glucose | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
  nmol/L.
Coefficient of variation (CV) of glucose measurements | From time of first unblinded CGM measurement (week 2) until time of last unblinded CGM measurement (week 12)
Participant with at least 70% heart rate (pulse) data (Yes/No) | From time of first heart rate measurement (week 0) until 12 weeks after the time of first heart rate measurement
  Count of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Digital/virtual site, Copenhegan, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com